CLINICAL TRIAL: NCT04164823
Title: The Effect of Taping in Reducing the Intensity of Pain in Primary Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Elena Estebanez de Miguel, Principal Investigator, Universidad de Zaragoza
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PI17/157
Record Dates: First submitted 2019-11-12; First posted 2019-11-15 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Primary Dysmenorrhea
Keywords: Primary Dysmenorrhea; Taping; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medical Taping (Experimental): Medical taping will be applied as a self-treatment. All participants will be instructed in an indvidual session and will receive a tutorial video to remember the kinesiotaping procedure. 3 band of a special and hypoallergenic tape (Kinematix Tex) will be attached to the abdominal (2 strips) and lower back (1 strip).
  Patients will be taped for four days. It will start at the beginning of pain associated to the menstruation.
  Interventions: Device: Medical taping
- Analgesic self-medication (OTC) (Active Comparator): Participants will use the usual analgesic self-treatment for primary dysmenorrhea.It will start at the beginning of pain associated to the menstruation.
  They will note the treatment indicating the analgesic and the dosage in a calendar.
  Interventions: Drug: Analgesic self-medication (OTC)

INTERVENTIONS:
Device: Medical taping — For the medical taping group, a piece of Kinesio tape 5 cm in width and 7-8 cm in length will be applied right from below the navel and will reach to where the pubic hair begins, and another piece of tape 10 cm in length will be applied to make a cross shape with the first piece. A tape of 20cm in length will be placed horizontally to the lower back.
  Arms: Medical Taping
Drug: Analgesic self-medication (OTC) — Participants will note the usual analgesic self-medication used to relief pain (ibuprofen, acetaminophen...).
  Arms: Analgesic self-medication (OTC)

SUMMARY:
To determine the effectiveness of kinesiotaping on pain in primary dysmenorrhea

DETAILED DESCRIPTION:
Primary dysmenorrhea is defined as cramping pain in the lower abdomen occurring just before or during menstruation, in the absence of other diseases.

About 50-90% of the women experience menstrual pain, and approximately 15% of them suffer from a severe level of pain It is a common cause of absenteeism and reduced quality of life in women.

From 21% to 96% of women with menstrual pain, reported to practice self-treatment either by pharmacological or nonpharmacological interventions. However, there are adverse events associated with the use of these drugs, including stomach ache, diarrhea, nausea, cutaneous reactions, liver or kidney damage or cardiovascular risk after discontinuing medication . Therefore, many patients with menstrual pain usually seek complementary and alternative techniques.

Medical taping concept is an alternative treatment that use elastic adhesive tape, which is applied to the patient's skin under tension.

It has the characteristic to cause elevation of the epidermis and thereby reduce the pressure on the mechanoreceptors below the dermis. This would have the effect of reducing nociceptive stimuli.

ELIGIBILITY:
Inclusion Criteria:

* Women presenting menstrual pain, 4 or more in VAS.
* Have attended gynecological examination in the past 18 months and had ever diagnosed as having a gynecological disorder different from primary dysmenorrhea
* Not have been diagnosed with secondary dysmenorrhea
* Regular menstrual cycles (cycle typical range of 21 to 35 days)
* Do not use an intrauterine contraceptive device (IUD) or taking oral contraceptive pills
* Nulliparous
* Ability to complete questionnaires in Spanish.

Exclusion Criteria:

* Women with mild dysmenorrhea (pain lower 4 in a numeric pain scale range 0-10);
* Women with irregular or infrequent menstrual cycles (outside the typical range of cycle 21 to 35 days);
* Women using an intrauterine contraceptive device (IUD) or taking oral contraceptive pills.
* Women who suffer from diseases diagnosed added
* Women to which it has undergone a surgical procedure for the treatment
* Provide skin lesions in the abdominal wall or in lumbar region
* Use or abuse of drugs or alcohol

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Change in menstrual pain with Visual Analogic Scale (VAS) | Participants will be followed for 6 menstrual cycles. Evaluations will be performed before, and just after 2 hours, 8 hours, 12 hours, 24 hours, and 48 hours after treatment in each menstrual cycle.
  VAS is a method of representing subjects' pain on a 10 cm linear scale. In this study, a score of 0 means 'a very low degree of pain' and 10 means 'a very high degree of pain

SECONDARY OUTCOMES:
Patient satisfaction with Visual Analogic Scale (VAS) | Participants will be followed for 6 menstrual cycles. Evaluations will be performed at the end of each treatment, when menstrual pain disappears (4-5 days after the beginning of the menstrual bleeding).
  Participants will note the self-care applied to relief menstrual pain indicating the VAS is a method of representing subjects' satisfaction with treatment on a 10 cm linear scale. In this study, a score of 0 means 'a very low degree of satisfaction with treatment' and 10 means 'a very high degree of satisfaction with treatment

CONTACTS AND LOCATIONS:
Overall Officials: Elena Estébanez de Miguel, Study Director — Universidad de Zaragoza
Locations (1):
- Elena Estébanez de Miguel, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lu Z, Li X, Chen R, Guo C. Kinesio taping improves pain and function in patients with knee osteoarthritis: A meta-analysis of randomized controlled trials. Int J Surg. 2018 Nov;59:27-35. doi: 10.1016/j.ijsu.2018.09.015. Epub 2018 Sep 28. PMID 30273684
- [Background] Macedo LB, Richards J, Borges DT, Melo SA, Brasileiro JS. Kinesio Taping reduces pain and improves disability in low back pain patients: a randomised controlled trial. Physiotherapy. 2019 Mar;105(1):65-75. doi: 10.1016/j.physio.2018.07.005. Epub 2018 Jul 26. PMID 30348455
- [Background] Espi-Lopez GV, Ingles M, Ferrando AC, Serra-Ano P. Effect of Kinesio taping on clinical symptoms in people with fibromyalgia: A randomized clinical trial. J Back Musculoskelet Rehabil. 2019;32(4):561-567. doi: 10.3233/BMR-171100. PMID 30530959
- [Background] Choi JH. Effects of kinesio taping and hot packs on premenstrual syndrome in females. J Phys Ther Sci. 2017 Sep;29(9):1514-1517. doi: 10.1589/jpts.29.1514. Epub 2017 Sep 15. PMID 28931978
- [Background] Campbell MA, McGrath PJ. Use of medication by adolescents for the management of menstrual discomfort. Arch Pediatr Adolesc Med. 1997 Sep;151(9):905-13. doi: 10.1001/archpedi.1997.02170460043007. PMID 9308868
- [Background] Grandi G, Ferrari S, Xholli A, Cannoletta M, Palma F, Romani C, Volpe A, Cagnacci A. Prevalence of menstrual pain in young women: what is dysmenorrhea? J Pain Res. 2012;5:169-74. doi: 10.2147/JPR.S30602. Epub 2012 Jun 20. PMID 22792003
- [Background] O'Connell K, Davis AR, Westhoff C. Self-treatment patterns among adolescent girls with dysmenorrhea. J Pediatr Adolesc Gynecol. 2006 Aug;19(4):285-9. doi: 10.1016/j.jpag.2006.05.004. PMID 16873033